CLINICAL TRIAL: NCT01943877
Title: Propolis In The Treatment Of Chronic Periodontitis - A Clinicomicrobiologic Study
Brief Title: Propolis In The Treatment Of Periodontitis
Acronym: PROPOLIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rajarajeswari Dental College & Hospital (Other)
Responsible Party: Principal Investigator, NEHAL N SANGHANI, mds, DR., Rajarajeswari Dental College & Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 971987
Record Dates: First submitted 2013-09-02; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Propolis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propolis (Experimental)
  Interventions: Procedure: scaling root planing; Drug: Propolis
- scaling and root planing (Sham Comparator)
  Interventions: Procedure: scaling root planing

INTERVENTIONS:
Procedure: scaling root planing — scaling root planing
Drug: Propolis — experimental
  Arms: Propolis

SUMMARY:
This study was conducted to evaluate by clinical and microbiological parameters the effect of locally delivered propolis as an adjunct to scaling and root planing in the treatment of chronic periodontitis.

DETAILED DESCRIPTION:
Materials and Methods: 20 subjects diagnosed with chronic periodontitis were recruited to participate in split-mouth design and provided informed consent. Subgingival plaque sampling and clinical recording at baseline, 15 days and 1 month was performed. The patients received scaling and root planing, followed by Propolis administration subgingivally in the test sites. Significant differences between test and control were evaluated using the Mann-Whitney U test and Wilcoxon rank test.

ELIGIBILITY:
Inclusion Criteria:

* good general health
* chronic periodontitis
* minimum of 20 natural teeth with at least one pocket per quadrant
* probing depth (PD) between 5 and 8 mm.

Exclusion Criteria:

* subgingival instrumentation within 3 months
* antibiotic therapy within 3 months prior to the start of the study;
* smokers
* pregnant or nursing women
* intolerance or allergy to honey products

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Change in the probing pocket depth and clinical attachment level | three time points of baseline,2 weeks, 4 weeks

SECONDARY OUTCOMES:
change in gingival index and microbiological changes | three time points baseline, 2 weeks, 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Rajarajeswari Dental College and Hospital, Bangalore, Karnataka, India